CLINICAL TRIAL: NCT06387719
Title: Precursors of Binge Eating Disorder in a Clinical Sample of Adolescents With Obesity: Early MRI Markers of Brain Reward and Inhibition Processing Dysfunction
Brief Title: Precursors of Binge Eating Disorder in a Clinical Sample of Adolescents With Obesity
Acronym: PREC-BED
Status: Recruiting | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: PREC-BED Study
Record Dates: First submitted 2024-02-27; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Binge-Eating Disorder; Obesity; Eating Disorders; BED; Other Specified Feeding or Eating Disorder; Eating Disorder Nos; Emotion Regulation; Food Addiction
Keywords: Binge Eating Disorder; Mental Health; Adolescents; Loss of control; Emotional eating; BED; youths; neuroimaging; reward response; response inhibition; magnetic resonance
MeSH Terms: conditions — Binge-Eating Disorder; Obesity; Feeding and Eating Disorders; Emotional Regulation; Food Addiction; Psychological Well-Being; Emotional Eating | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Neuroimaging
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group (CG): Adolescents with obesity, measured as body mass index (BMI) z-score above 2 standard deviations, and no BED/PREC-BED
  Interventions: Diagnostic Test: Magnetic resonance imaging
- BED group: adolescents with obesity, measured as BMI z-score above 2 standard deviations, and BED
  Interventions: Diagnostic Test: Magnetic resonance imaging
- PREC-BED group: adolescents with obesity, measured as BMI z-score above 2 standard deviations, PREC-BED
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — * Basic sequence for ethical consideration: evaluation of casual findings.
  * Structural MRI.
  * Functional MRI (fMRI) in the Resting-state
  * fMRI- task based. Presented in a computer screen on a magnetically compatible googles.
  Other Names: Clinical assessment; Neurocognitive assessment

SUMMARY:
BACKGROUND: Binge eating disorder (BED) is the worldwide most-prevalent eating disorder. It is associated with psychiatric comorbidities and obesity, a high impact in life functioning, and high morbidity and mortality. First symptoms appear frequently in youths, who most commonly present incomplete (subthreshold) criteria for BED (precursor forms, PREC-BED). While some subjects will evolve from PREC-BED to BED, there is no gold standard to identify the clinical evolution. Information from prior studies suggest early alterations in reward and inhibitory brain circuits in PREC-BED may predict increased vulnerability or resilience to develop BED. Tools based on MRI brain connectivity analyses (MRI-BC), built on robust and interpretable connectivity whole-brain models, have proven successful in diagnostic classification and predicting certain clinical outcomes. OBJECTIVES: To study MRI-BC diagnostic markers of PREC-BED and to explore prognosis at 1 year of follow-up in a sample of adolescents with obesity (12-17 years old). METHODS: A) Transversal analytical design: 3-group (n=34 per group) comparison of neuroimaging (MRI-BC), neurocognitive and clinical markers in adolescents with obesity and i) BED, ii) PREC-BED, iii) no BED nor PREC-BED (Healthy group, HC). B) Longitudinal analytical design, pilot, exploratory: adolescents with PREC-BED will be evaluated in clinical and neurocognitive variables at 1 year. Baseline brain neuroimaging variables (alone and in combination with clinical and neurocognitive variables) will be analyzed as predictors of clinical prognosis, including conversion to BED.

DETAILED DESCRIPTION:
Background

Binge eating disorder (BED) has been a diagnosis on its own only since the last edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) in 2013. It is the most prevalent eating disorder worldwide, affecting more than 50 million subjects, world-wide. BED is characterized by binge eating episodes: eating a large amount of food in a discrete period and with a sense of lack of control. Two main peaks of onset have been identified: one is at mean age 14 and the second between 18-20 years old. BED is one of the primary chronic illnesses among adolescents and is commonly associated with psychiatric comorbidities (more than 60% of lifetime prevalence), but also with obesity and its physical consequences, showing a high impact in life functioning and a high morbi-mortality. BED prevalence in youth populations is between 1-3%, and up to 37% in adolescent population with obesity. These figures have raised in parallel with the high increase in obesity prevalence in this population. When considering subclinical presentations in the general population, which involve presenting some symptoms but not fulfilling all the diagnostic criteria for BED, the prevalence is 3%. Subclinical forms are described with terms such as emotional eating, disorganized eating, loss of control eating, among others. The latter is the only construct that has operationalized criteria. In some cases, but not all, individuals with these conditions might be diagnosed with specified or unspecified DSM-5 eating disorder categories ("other specified feeding or eating disorder" -OSFED-, or "eating disorder not otherwise specified" -EDNOS-).

The first symptoms of BED often appear in youths, who frequently exhibit incomplete criteria, which are associated with a future development of BED (i.e. subclinical forms or precursor forms, PREC-BED). These subclinical forms are more frequent in adolescents, in comparison to adults. The factors determining the conversion from PREC-BED to BED are unknown and to our knowledge, only one study evaluated the percentage of conversion to BED in a small sample of adolescents with PREC-BED, finding a 28% conversion rate. There is no gold standard for identifying the clinical progression of incomplete forms, which hinders prevention and personalized treatment.

The most kown underlying factor identified in BED is a dysfunction in emotional regulation, and neuroimaging studies have identified alterations in relevant brain circuits involved in these functions, such as reward response and response inhibition. These alterations are observed in BED and seem to be present in PREC-BED and could potentially predict a greater vulnerability or resilience to developing BED in the future. For example: Reward response: Subjects with BED present increased preference for immediate reward (as opposed to delayed), greater food-reward sensitivity and greater rash-spontaneous behaviour in the context of food. At the brain level, despite the scarce evidence, a large longitudinal study (i.e. Adolescent Brain Cognitive Development -ABCD- study) suggests that early brain structural differences during childhood of key reward regions (i.e. nucleus accumbens) might be a genetic predisposition for the development of obesity and possibly of an altered pattern of eating. In adult samples of BED, a few studies found structural or functional alterations in regions of the reward system. Inhibition: Evidences of poor impulse control or decreased inhibitory control come from adult samples, but also from the limited samples in youth, which are also limited. In adolescents with PREC-BED, some studies found hypoactivations during inhibitory processing regions, or during the inhibition of emotions in the the context of negative mood induction through a peer interaction paradigm. In another study, hyperactivations (as opposite to hypoactivations) of self-regulatory regions when receiving milkshake flavours during the neuroimaging session, were suggested as compensatory early mechanisms, representing an increased cognitive effort to regulate emotions under such restrictive conditions. Studies in BED were only found in adults.

Neuroimaging techniques using magnetic resonance imaging (MRI) allow for non-invasive study of live brain activity, which can be done during the participation of the subject in a task (for example, an inhibition task or a response processing task). This would allow the visualization of functional deficits evidenced during a cognitive demand; in the same manner the cardiologist may realize exercise tolerance test. Advanced MRI techniques nowadays offer unique insights into the anatomical and functional architecture of the brain. For example, advanced MRI brain connectivity (MRI-BC) techniques incorporate the modelling of brain dynamics between regions, which approximates to the inherent complexity of brain architecture and psychiatric disorders and open new perspective to investigate circuits and alterations involved in neurological and diseases. Such analysis can be conducted during a resting state in the MRI session, but also during specific task (for example, inhibition response task or reward-based task). One of the available whole-brain models of MRI-BC is called effective connectivity (EC), which provides information of the hierarchical or directional connectivity and/or activation between brain regions and networks. Our team (UPF team members) has developed a new technique to estimate EC, the MOU-EC generative model (Multivariate Ornstein-Uhlenbeck), which improves interpretability over other techniques and has been shown its relevance in predicting outcomes. Similar advanced techniques have proven useful in a few studies in eating disorders, including children with BED in one study and in EC in taste and food intake regulating circuits in anorexia and bulimia nervosa.

The development of prognostic markers in PREC-BED forms in the child and adolescent population would be highly relevant to increase the detection of these forms, prevent the development of BED, and enable early and personalized treatment. While neuroimaging markers alone and for diagnostic purposes have not yielded the expected results in other pathologies, it is possible that MRI-BC alone or in combination with other clinical and neuropsychological variables could constitute more sensitive and specific predictive models of risk, especially in pathologies with a bio-psychosocial origin like BED.

PROJECT'S AIM

The aim is to characterize regulation (reward and inhibition-based) processes in PREC-BED and BED in adolescents and to explore MRI-BC neurobiological markers of PREC-BED diagnosis and of prognosis at 1 year of follow-up.

FUNDING

Grant by the Instituto de Salud Carlos III (Ministerio de Ciencia, Innovación y Universades) and the private company Torrons Vicens.

ELIGIBILITY:
Inclusion Criteria:

* Patients derived to the Endocrinology Department with obesity as the main criterion for consultation, measured as body mass index (BMI) z-score above 2 standard deviations.
* Age between 12-16 years old.
* Signed informed consent by parents or legal guardians of subjects, plus the signed consent by the adolescent when being 12 or older years/old.

Additional inclusion criteria for the BED and PREC-BED groups:

* The presence of DSM-5 criteria for BED in the BED group.
* Fulfilling the LOC (loss of control) criteria (related to the original Marcus&Kalarchian) in the PREC-BED group.

Exclusion Criteria:

* Intelligence quotient < 70 measured with the K-BIT.
* Any comorbid psychiatric disorder, except BED in the BED group or PREC-BED in the PREC-BED group. Tobacco use and the presence of an adaptative disorder or any mild anxiety disorder will be accepted in all groups.
* Traumatic brain injury or any neurological disorder.
* Use of dental braces (due to important artifact in MRI).
* MRI: Absolute contraindications (e.g.: metal objects), relative contraindications (claustrophobia). Anthropometric measures: Weight > 150Kg or shoulder to shoulder measurement > 70 cm.
* Any severe medical conditions (including Sleep apnea-hypopnea syndrome), except for obesity and metabolic syndrome.
* Not signing the informed consent.
* Pregnancy for females.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents with obesity (12-16 y/o) would be consecutively asked to participate when attending their visits at the Endocrinology Department at Hospital Sant Joan de Déu (HSJD).
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging assessment | Baseline (transversal design)
  Connectivity analyses using Effective-connectivity (EC) in whole-brain models
Neuroimaging assessment | Baseline (transversal design)
  Brain response during task-based fMRI (Monetary incentive Delay Task, Stop Signal task)

SECONDARY OUTCOMES:
Height | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Height in centimeters
Weight | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Weight in kilograms
Waist perimeter | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Waist perimeter in centimeters
BMI | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Weight and height will be combined to report BMI in kg/m^2
Blood pressure | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Blood pressure in mm Hg
Fasting glucose | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Fasting glucose in mg/dl
Triglycerides | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Triglycerides in mg/dl
HDL cholesterol | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  HDL cholesterol in mg/dl
Developmental Tanner stage | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  The scale defines physical measurements of development based on external primary and secondary sex characteristics.
Adherence to Mediterranean diet | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  Self-administered questionnaire (The Kid-MED). Units on a Scale: Total score from 0 to 12. Score ≥8: Optimal dietary quality.
  Score 4-7: Intermediate dietary quality. Improvements are needed to enhance adherence to the MedDiet.
  Score ≤3: Very low dietary quality.
Diagnosis of BED, and PREC-BED or exclusion of other DMS-5 diagnosis. | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  The Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS-PL): semi-structured interview to parents or legal guardians and subjects aimed to diagnosis mental disorders based on DMS-5 criteria, administered by health care providers (clinician).
Functioning | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  Global Assessment of Functioning (GAF) Scale (clinician). Units on a scale: 11 to 100, higher scores will indicate a better outcome.
Depression | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  Beck Depression Inventory for Children (BYI-2): Spanish adapted self-administered questionnaire for depressive symptoms (child)
  T-scores:
  * ≥70 Very high
  * 60-69 Quite high
  * 55-59 Somewhat high
  * <55 Average
Anxiety | Baseline and 1-year follow-up (for the HG and PREC-BED groups).
  The Screen for Child Anxiety Related Disorders (SCARED). A total score of 25 may indicate the presence of an anxiety disorder. Scores higher than 30 are more specific.
Emotion Regulation | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  Difficulties Emotion Regulation Scale (DERS): Subscales and total scores are obtained by the sum of the corresponding items and higher scores indicate more difficulties in Emotional Regulation.
Eating symptomatology | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  Eating Disorder Examination Questionnaire-Adolescents (EDE-Q-A): It generates three scales a) the Restraint subscale, b) the Weight, Figure and Eating Concern subscale, and c) the Total scale. Higher scores mean a worse outcome.
Eating symptomatology | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  - Emotional Eating Scale Adapted for Children and Adolescents (EES-C): It generates subscales (anger, anxiety, depression, restlessness and hopelessness). higher scores mean a worse outcome
Temperamental tendencies for sensitivity to punishment and sensitivity to reward. | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  The Sensitivity to Punishment and Sensitivity to Reward Questionnaire Junior (SPSRQ-J). It generates two subscales sensitivity to punishment and sensitivity to reward.
Food Addiction | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  Yale Food Addiction Scale for Children (YFAS-C): The scores provide an assessment of food addiction in two different ways. On one hand, the "symptom count," which offers a scoring version reflecting the number of dependency symptoms based on the 7 described criteria without considering clinical importance in the scoring (minimum 0, maximum 7 points). And, on the other hand, the "addiction diagnosis," which evaluates whether the diagnosis of food addiction can be established or not, and is confirmed when there are three or more symptoms present and significant clinical distress or impairment (questions 15 and 16).
Food intake | Baseline and 1-year follow-up (for the HG and PREC-BED groups)
  Questionnaire on frequency of dietary intake (CFCA): The NOVA classification will be used to extract information of the intake of ultra-processed foods and drinks for each subject (daily grams of UPFD intake/total daily grams, multiplied by 100) for each participant (world.openfoodfacts.org).
General Intelligence | Baseline
  Kaufman Brief Intelligence Test (K-BIT): Standard scores have a mean of 100 and a standard deviation of 15
Attention ability | Baseline
  Continuous Performance Test (CPT-IP). T-score: The values of the scores depend on the variables.
Visuo-constructional ability and visual memory | Baseline
  Rey-Osterrieth complex figures task. Standardized scores: higher scores mean a better outcome.
Executive function: cognitive flexibility, alternating attention, sequencing, visual search, and motor speed. | Baseline.
  Trail Making Test (TMT). Standardized scores: higher scores mean a better outcome.
Executive function: working memory ability | Baseline.
  Letter-number sequencing (subtest of the Wechsler Intelligence Scale for Children-Fifth Edition - WISC-V).
  Standardized scores: higher scores mean a better outcome.
Executive function: decision-making abilities reward based | Baseline.
  Iowa gambling task Standardized scores: higher scores mean a better outcome.
Executive function: ability to inhibit cognitive interference | Baseline.
  Stroop Test. Standardized scores: higher scores mean a better outcome.
Executive function: planning and strategic organisation | Baseline.
  Rey-Osterrieth complex figures task. Standardized scores: higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Via, PhD, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual deidentified participant data may be provided to qualified researchers with academic interest in eating disorders. Data shared will be pseudonymised, with no Protected Health Information (PHI included).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Proposals should be directed to the principal investigator. To gain access, data requestors will need to sign a data agreement with our institution, to comply with legal requirements and data protection rights. The study protocol and/or an amendment to the protocol will be reviewed by the corresponding Ethics Committees.

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders (5th Ed.). Washington, DC; 2013.
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders. American Psychiatric Association; 2013. doi:10.1176/appi.books.9780890425596
- [Background] Erskine HE, Whiteford HA. Epidemiology of binge eating disorder. Curr Opin Psychiatry. 2018 Nov;31(6):462-470. doi: 10.1097/YCO.0000000000000449. PMID 30113324
- [Background] Santomauro DF, Melen S, Mitchison D, Vos T, Whiteford H, Ferrari AJ. The hidden burden of eating disorders: an extension of estimates from the Global Burden of Disease Study 2019. Lancet Psychiatry. 2021 Apr;8(4):320-328. doi: 10.1016/S2215-0366(21)00040-7. Epub 2021 Mar 3. PMID 33675688
- [Background] Vannucci A, Nelson EE, Bongiorno DM, Pine DS, Yanovski JA, Tanofsky-Kraff M. Behavioral and neurodevelopmental precursors to binge-type eating disorders: support for the role of negative valence systems. Psychol Med. 2015 Oct;45(14):2921-36. doi: 10.1017/S003329171500104X. Epub 2015 Jun 4. PMID 26040923
- [Background] American Psychiatric Association. Anxiety Disorders. In: Diagnostic and Statistical Manual of Mental Disorders. American Psychiatric Association; 2013. doi:10.1176/appi.books.9780890425596.dsm05
- [Background] Marzilli E, Cerniglia L, Cimino S. A narrative review of binge eating disorder in adolescence: prevalence, impact, and psychological treatment strategies. Adolesc Health Med Ther. 2018 Jan 5;9:17-30. doi: 10.2147/AHMT.S148050. eCollection 2018. PMID 29379325
- [Background] Guerdjikova AI, Mori N, Casuto LS, McElroy SL. Update on Binge Eating Disorder. Med Clin North Am. 2019 Jul;103(4):669-680. doi: 10.1016/j.mcna.2019.02.003. PMID 31078199
- [Background] van Wijnen LG, Boluijt PR, Hoeven-Mulder HB, Bemelmans WJ, Wendel-Vos GC. Weight status, psychological health, suicidal thoughts, and suicide attempts in Dutch adolescents: results from the 2003 E-MOVO project. Obesity (Silver Spring). 2010 May;18(5):1059-61. doi: 10.1038/oby.2009.334. Epub 2009 Oct 8. PMID 19834472
- [Background] Smink FR, van Hoeken D, Oldehinkel AJ, Hoek HW. Prevalence and severity of DSM-5 eating disorders in a community cohort of adolescents. Int J Eat Disord. 2014 Sep;47(6):610-9. doi: 10.1002/eat.22316. Epub 2014 Jun 5. PMID 24903034
- [Background] Tanofsky-Kraff M, Marcus MD, Yanovski SZ, Yanovski JA. Loss of control eating disorder in children age 12 years and younger: proposed research criteria. Eat Behav. 2008 Aug;9(3):360-5. doi: 10.1016/j.eatbeh.2008.03.002. Epub 2008 Apr 7. PMID 18549996
- [Background] Decaluwe V, Braet C. Prevalence of binge-eating disorder in obese children and adolescents seeking weight-loss treatment. Int J Obes Relat Metab Disord. 2003 Mar;27(3):404-9. doi: 10.1038/sj.ijo.0802233. PMID 12629570
- [Background] Mitchison D, Touyz S, Gonzalez-Chica DA, Stocks N, Hay P. How abnormal is binge eating? 18-Year time trends in population prevalence and burden. Acta Psychiatr Scand. 2017 Aug;136(2):147-155. doi: 10.1111/acps.12735. Epub 2017 Apr 16. PMID 28419425
- [Background] Kjeldbjerg ML, Clausen L. Prevalence of binge-eating disorder among children and adolescents: a systematic review and meta-analysis. Eur Child Adolesc Psychiatry. 2023 Apr;32(4):549-574. doi: 10.1007/s00787-021-01850-2. Epub 2021 Jul 27. PMID 34318368
- [Background] Tanofsky-Kraff M, Shomaker LB, Olsen C, Roza CA, Wolkoff LE, Columbo KM, Raciti G, Zocca JM, Wilfley DE, Yanovski SZ, Yanovski JA. A prospective study of pediatric loss of control eating and psychological outcomes. J Abnorm Psychol. 2011 Feb;120(1):108-18. doi: 10.1037/a0021406. PMID 21114355
- [Background] Neumark-Sztainer D, Wall M, Guo J, Story M, Haines J, Eisenberg M. Obesity, disordered eating, and eating disorders in a longitudinal study of adolescents: how do dieters fare 5 years later? J Am Diet Assoc. 2006 Apr;106(4):559-68. doi: 10.1016/j.jada.2006.01.003. PMID 16567152
- [Background] Vainik U, Neseliler S, Konstabel K, Fellows LK, Dagher A. Eating traits questionnaires as a continuum of a single concept. Uncontrolled eating. Appetite. 2015 Jul;90:229-39. doi: 10.1016/j.appet.2015.03.004. Epub 2015 Mar 10. PMID 25769975
- [Background] Hebebrand J, Gearhardt AN. The concept of "food addiction" helps inform the understanding of overeating and obesity: NO. Am J Clin Nutr. 2021 Feb 2;113(2):268-273. doi: 10.1093/ajcn/nqaa344. PMID 33448280
- [Background] Eldredge KL, Agras WS. Weight and shape overconcern and emotional eating in binge eating disorder. Int J Eat Disord. 1996 Jan;19(1):73-82. doi: 10.1002/(SICI)1098-108X(199601)19:13.0.CO;2-T. PMID 8640205
- [Background] Balantekin KN, Birch LL, Savage JS. Eating in the absence of hunger during childhood predicts self-reported binge eating in adolescence. Eat Behav. 2017 Jan;24:7-10. doi: 10.1016/j.eatbeh.2016.11.003. Epub 2016 Nov 10. PMID 27851989
- [Background] Herle M, Stavola B, Hubel C, Abdulkadir M, Ferreira DS, Loos RJF, Bryant-Waugh R, Bulik CM, Micali N. A longitudinal study of eating behaviours in childhood and later eating disorder behaviours and diagnoses. Br J Psychiatry. 2020 Feb;216(2):113-119. doi: 10.1192/bjp.2019.174. PMID 31378207
- [Background] Stice E, Marti CN, Rohde P. Prevalence, incidence, impairment, and course of the proposed DSM-5 eating disorder diagnoses in an 8-year prospective community study of young women. J Abnorm Psychol. 2013 May;122(2):445-57. doi: 10.1037/a0030679. Epub 2012 Nov 12. PMID 23148784
- [Background] Wierenga CE, Ely A, Bischoff-Grethe A, Bailer UF, Simmons AN, Kaye WH. Are Extremes of Consumption in Eating Disorders Related to an Altered Balance between Reward and Inhibition? Front Behav Neurosci. 2014 Dec 9;8:410. doi: 10.3389/fnbeh.2014.00410. eCollection 2014. PMID 25538579
- [Background] Treasure J, Duarte TA, Schmidt U. Eating disorders. Lancet. 2020 Mar 14;395(10227):899-911. doi: 10.1016/S0140-6736(20)30059-3. PMID 32171414
- [Background] Giel KE, Teufel M, Junne F, Zipfel S, Schag K. Food-Related Impulsivity in Obesity and Binge Eating Disorder-A Systematic Update of the Evidence. Nutrients. 2017 Oct 27;9(11):1170. doi: 10.3390/nu9111170. PMID 29077027
- [Background] Rapuano KM, Laurent JS, Hagler DJ Jr, Hatton SN, Thompson WK, Jernigan TL, Dale AM, Casey BJ, Watts R. Nucleus accumbens cytoarchitecture predicts weight gain in children. Proc Natl Acad Sci U S A. 2020 Oct 27;117(43):26977-26984. doi: 10.1073/pnas.2007918117. Epub 2020 Oct 12. PMID 33046629
- [Background] Donnelly B, Touyz S, Hay P, Burton A, Russell J, Caterson I. Neuroimaging in bulimia nervosa and binge eating disorder: a systematic review. J Eat Disord. 2018 Feb 20;6:3. doi: 10.1186/s40337-018-0187-1. eCollection 2018. PMID 29468065
- [Background] Aviram-Friedman R, Astbury N, Ochner CN, Contento I, Geliebter A. Neurobiological evidence for attention bias to food, emotional dysregulation, disinhibition and deficient somatosensory awareness in obesity with binge eating disorder. Physiol Behav. 2018 Feb 1;184:122-128. doi: 10.1016/j.physbeh.2017.11.003. Epub 2017 Nov 8. PMID 29128522
- [Background] Hagan KE, Bohon C. Subcortical brain volume and cortical thickness in adolescent girls and women with binge eating. Int J Eat Disord. 2021 Aug;54(8):1527-1536. doi: 10.1002/eat.23563. Epub 2021 Jun 1. PMID 34061404
- [Background] Turan S, Sarioglu FC, Erbas IM, Cavusoglu B, Karagoz E, Sisman AR, Guney SA, Guleryuz H, Abaci A, Ozturk Y, Akay AP. Altered regional grey matter volume and appetite-related hormone levels in adolescent obesity with or without binge-eating disorder. Eat Weight Disord. 2021 Dec;26(8):2555-2562. doi: 10.1007/s40519-021-01117-4. Epub 2021 Feb 6. PMID 33548051
- [Background] Bodell LP, Wildes JE, Goldschmidt AB, Lepage R, Keenan KE, Guyer AE, Hipwell AE, Stepp SD, Forbes EE. Associations Between Neural Reward Processing and Binge Eating Among Adolescent Girls. J Adolesc Health. 2018 Jan;62(1):107-113. doi: 10.1016/j.jadohealth.2017.08.006. Epub 2017 Oct 17. PMID 29054735
- [Background] Lavagnino L, Arnone D, Cao B, Soares JC, Selvaraj S. Inhibitory control in obesity and binge eating disorder: A systematic review and meta-analysis of neurocognitive and neuroimaging studies. Neurosci Biobehav Rev. 2016 Sep;68:714-726. doi: 10.1016/j.neubiorev.2016.06.041. Epub 2016 Jul 2. PMID 27381956
- [Background] Hardee JE, Phaneuf C, Cope L, Zucker R, Gearhardt A, Heitzeg M. Neural correlates of inhibitory control in youth with symptoms of food addiction. Appetite. 2020 May 1;148:104578. doi: 10.1016/j.appet.2019.104578. Epub 2020 Jan 2. PMID 31904390
- [Background] Jarcho JM, Tanofsky-Kraff M, Nelson EE, Engel SG, Vannucci A, Field SE, Romer AL, Hannallah L, Brady SM, Demidowich AP, Shomaker LB, Courville AB, Pine DS, Yanovski JA. Neural activation during anticipated peer evaluation and laboratory meal intake in overweight girls with and without loss of control eating. Neuroimage. 2015 Mar;108:343-53. doi: 10.1016/j.neuroimage.2014.12.054. Epub 2014 Dec 27. PMID 25550068
- [Background] Goldschmidt AB, Dickstein DP, MacNamara AE, Phan KL, O'Brien S, Le Grange D, Fisher JO, Keedy S. A Pilot Study of Neural Correlates of Loss of Control Eating in Children With Overweight/Obesity: Probing Intermittent Access to Food as a Means of Eliciting Disinhibited Eating. J Pediatr Psychol. 2018 Sep 1;43(8):846-855. doi: 10.1093/jpepsy/jsy009. PMID 29462339
- [Background] Xue G, Chen C, Lu ZL, Dong Q. Brain Imaging Techniques and Their Applications in Decision-Making Research. Xin Li Xue Bao. 2010 Feb 3;42(1):120-137. doi: 10.3724/SP.J.1041.2010.00120. PMID 20376329
- [Background] Kobeleva X, Varoquaux G, Dagher A, Adhikari M, Grefkes C, Gilson M. Advancing brain network models to reconcile functional neuroimaging and clinical research. Neuroimage Clin. 2022;36:103262. doi: 10.1016/j.nicl.2022.103262. Epub 2022 Nov 7. PMID 36451365
- [Background] Rolls ET, Cheng W, Gilson M, Gong W, Deco G, Lo CZ, Yang AC, Tsai SJ, Liu ME, Lin CP, Feng J. Beyond the disconnectivity hypothesis of schizophrenia. Cereb Cortex. 2020 Mar 14;30(3):1213-1233. doi: 10.1093/cercor/bhz161. PMID 31381086
- [Background] Adhikari MH, Griffis J, Siegel JS, Thiebaut de Schotten M, Deco G, Instabato A, Gilson M, Corbetta M. Effective connectivity extracts clinically relevant prognostic information from resting state activity in stroke. Brain Commun. 2021 Oct 23;3(4):fcab233. doi: 10.1093/braincomms/fcab233. eCollection 2021. PMID 34729479
- [Background] Murray SB, Alba C, Duval CJ, Nagata JM, Cabeen RP, Lee DJ, Toga AW, Siegel SJ, Jann K. Aberrant functional connectivity between reward and inhibitory control networks in pre-adolescent binge eating disorder. Psychol Med. 2023 Jul;53(9):3869-3878. doi: 10.1017/S0033291722000514. Epub 2022 Mar 18. PMID 35301976
- [Background] Frank GK, Shott ME, Riederer J, Pryor TL. Altered structural and effective connectivity in anorexia and bulimia nervosa in circuits that regulate energy and reward homeostasis. Transl Psychiatry. 2016 Nov 1;6(11):e932. doi: 10.1038/tp.2016.199. PMID 27801897
- [Background] Chamay-Weber C, Combescure C, Lanza L, Carrard I, Haller DM. Screening Obese Adolescents for Binge Eating Disorder in Primary Care: The Adolescent Binge Eating Scale. J Pediatr. 2017 Jun;185:68-72.e1. doi: 10.1016/j.jpeds.2017.02.038. Epub 2017 Mar 10. PMID 28285753
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Endicott J, Spitzer RL, Fleiss JL, Cohen J. The global assessment scale. A procedure for measuring overall severity of psychiatric disturbance. Arch Gen Psychiatry. 1976 Jun;33(6):766-71. doi: 10.1001/archpsyc.1976.01770060086012. PMID 938196
- [Background] Beck JS, Beck AT, Jolly J, Steer RA, Assessment Library Materials (University of Lethbridge. Faculty of Education. Curriculum Laboratory). Beck Youth Inventories for Children and Adolescents : Manual. 2nd ed. PsychCorp; 2005.
- [Background] Dpto. I+D Pearson Clinical & Talent Assessment colaboración con Dña. Victoria del Barrio, D. José Pedro Espada, Dña. Eva España DñaAI y DñaMÁM. BYI-2 , Inventarios de Beck para niños y adolescentes-2 - Pearson Clinical & Talent Assessment. Accessed March 3, 2022. https://www.pearsonclinical.es/byi-2-inventarios-de-beck-para-ninos-y-adolescentes-2
- [Background] Forcadell E, Medrano L, Garcia-Delgar B, Fernandez-Martinez I, Orgiles M, Garcia C, Lazaro L, Lera-Miguel S. Psychometric Properties of the Children's Version of the Spence Children's Anxiety Scale (SCAS) in a Spanish Clinical Sample. Span J Psychol. 2020 Oct 20;23:e40. doi: 10.1017/SJP.2020.39. PMID 33079028
- [Background] Birmaher B, Khetarpal S, Brent D, Cully M, Balach L, Kaufman J, Neer SM. The Screen for Child Anxiety Related Emotional Disorders (SCARED): scale construction and psychometric characteristics. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):545-53. doi: 10.1097/00004583-199704000-00018. PMID 9100430
- [Background] Gratz KL, Roemer L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale 1. J Psychopathol Behav Assess. 2004;26(1).
- [Background] Hervás G, Jódar R. Adaptación al castellano de la Escala de Dificultades en la Regulación Emocional The spanish version of the Difficulties in Emotion Regulation Scale. 2008;19(2):139-156.
- [Background] Tanofsky-Kraff M, Theim KR, Yanovski SZ, Bassett AM, Burns NP, Ranzenhofer LM, Glasofer DR, Yanovski JA. Validation of the emotional eating scale adapted for use in children and adolescents (EES-C). Int J Eat Disord. 2007 Apr;40(3):232-40. doi: 10.1002/eat.20362. PMID 17262813
- [Background] Perpina C, Cebolla A, Botella C, Lurbe E, Torro MI. Emotional Eating Scale for children and adolescents: psychometric characteristics in a Spanish sample. J Clin Child Adolesc Psychol. 2011;40(3):424-33. doi: 10.1080/15374416.2011.563468. PMID 21534053
- [Background] Torrubia R, Avila C, Molto J, et al. The Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ) as a measure of Gray's anxiety and impulsivity dimensions. Pers Individ Dif. 2001;31(6):834-862. doi:10.1016/S0191-8869(00)00183-5
- [Background] Gearhardt AN, Roberto CA, Seamans MJ, Corbin WR, Brownell KD. Preliminary validation of the Yale Food Addiction Scale for children. Eat Behav. 2013 Dec;14(4):508-12. doi: 10.1016/j.eatbeh.2013.07.002. Epub 2013 Jul 21. PMID 24183146
- [Background] Benitez Brito N, Pinto Robayna B, Ramallo Farina Y, Moreno Redondo F, Leon Salas B, Diaz Romero C. [Cross-cultural validation of the Yale Food Addiction Scale for Children (YFAS-c) into the Spanish language to assess food addiction in the pediatric population]. Span J Psychiatry Ment Health. 2024 Oct-Dec;17(4):222-230. doi: 10.1016/j.rpsm.2021.11.006. Epub 2021 Nov 17. Spanish. PMID 39710879
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Sepulveda AR, Compte EJ, Faya M, Villasenor A, Gutierrez S, Andres P, Graell M. Spanish validation of the Eating Disorder Examination Questionnaire for Adolescents (EDE-Q-A): confirmatory factor analyses among a clinical sample. Eat Disord. 2019 Nov-Dec;27(6):565-576. doi: 10.1080/10640266.2019.1567154. Epub 2019 Feb 13. PMID 30758263
- [Background] Sysko R, Walsh BT, Fairburn CG. Eating Disorder Examination-Questionnaire as a measure of change in patients with bulimia nervosa. Int J Eat Disord. 2005 Mar;37(2):100-6. doi: 10.1002/eat.20078. PMID 15732070
- [Background] Rodriguez IT, Ballart JF, Pastor GC, Jorda EB, Val VA. [Validation of a short questionnaire on frequency of dietary intake: reproducibility and validity]. Nutr Hosp. 2008 May-Jun;23(3):242-52. Spanish. PMID 18560701
- [Background] Kaufman AS, Cordero Pando A, Calonge Isabel, Kaufman NL. K-BIT : test breve de inteligencia de Kaufman. Published online 2011.
- [Background] Conners CK, Sitarenios G. Conners' Continuous Performance Test (CPT). In: Encyclopedia of Clinical Neuropsychology. Springer New York; 2011:681-683. doi:10.1007/978-0-387-79948-3_1535
- [Background] Reitan RM. Trail Making Test. Manual for Administration, Scoring, and Interpretation. . : Indiana University Press.; 1956.
- [Background] Wechsler D. WISC-V, Escala de Inteligencia de Wechsler Para Niños-V - Pearson Clinical & Talent Assessment. (NCS Pearson Inc. (Pearson Assessment)., ed.).; 2014.
- [Background] Bechara A, Damasio AR, Damasio H, Anderson SW. Insensitivity to future consequences following damage to human prefrontal cortex. Cognition. 1994 Apr-Jun;50(1-3):7-15. doi: 10.1016/0010-0277(94)90018-3. PMID 8039375
- [Background] Golden CJ. A group version of the Stroop Color and Word Test. J Pers Assess. 1975 Aug;39(4):386-8. doi: 10.1207/s15327752jpa3904_10. PMID 16367401
- [Background] Silverman MH, Krueger RF, Iacono WG, Malone SM, Hunt RH, Thomas KM. Quantifying familial influences on brain activation during the monetary incentive delay task: an adolescent monozygotic twin study. Biol Psychol. 2014 Dec;103:7-14. doi: 10.1016/j.biopsycho.2014.07.016. Epub 2014 Aug 4. PMID 25101864
- [Background] Bartholdy S, O'Daly OG, Campbell IC, Banaschewski T, Barker G, Bokde ALW, Bromberg U, Buchel C, Quinlan EB, Desrivieres S, Flor H, Frouin V, Garavan H, Gowland P, Heinz A, Ittermann B, Martinot JL, Paillere Martinot ML, Nees F, Orfanos DP, Poustka L, Hohmann S, Frohner JH, Smolka MN, Walter H, Whelan R, Schumann G, Schmidt U; IMAGEN Consortium. Neural Correlates of Failed Inhibitory Control as an Early Marker of Disordered Eating in Adolescents. Biol Psychiatry. 2019 Jun 1;85(11):956-965. doi: 10.1016/j.biopsych.2019.01.027. Epub 2019 Mar 25. PMID 31122340
- [Background] Marcus MD, Kalarchian MA. Binge eating in children and adolescents. Int J Eat Disord. 2003;34 Suppl:S47-57. doi: 10.1002/eat.10205. PMID 12900986
- [Background] Shapiro JR, Woolson SL, Hamer RM, Kalarchian MA, Marcus MD, Bulik CM. Evaluating binge eating disorder in children: development of the children's binge eating disorder scale (C-BEDS). Int J Eat Disord. 2007 Jan;40(1):82-9. doi: 10.1002/eat.20318. PMID 16958120
- [Background] Cebolla A, Perpina C, Lurbe E, Alvarez-Pitti J, Botella C. [Prevalence of binge eating disorder among a clinical sample of obese children]. An Pediatr (Barc). 2012 Aug;77(2):98-102. doi: 10.1016/j.anpedi.2011.11.027. Epub 2012 Feb 10. Spanish. PMID 22326512
- [Background] Miranda-Olivos R, Steward T, Martinez-Zalacain I, Mestre-Bach G, Juaneda-Segui A, Jimenez-Murcia S, Fernandez-Formoso JA, Vilarrasa N, Veciana de Las Heras M, Custal N, Virgili N, Lopez-Urdiales R, Menchon JM, Granero R, Soriano-Mas C, Fernandez-Aranda F. The neural correlates of delay discounting in obesity and binge eating disorder. J Behav Addict. 2021 Apr 26;10(3):498-507. doi: 10.1556/2006.2021.00023. Print 2021 Oct 5. PMID 33950859
- [Background] Pallares V, Insabato A, Sanjuan A, Kuhn S, Mantini D, Deco G, Gilson M. Extracting orthogonal subject- and condition-specific signatures from fMRI data using whole-brain effective connectivity. Neuroimage. 2018 Sep;178:238-254. doi: 10.1016/j.neuroimage.2018.04.070. Epub 2018 May 22. PMID 29753842
- See also: Organization WH. Obesidad y sobrepeso. Published 2023. Accessed April 23, 2023. — http://www.who.int/es/news-room/fact-sheets/detail/obesity-and-overweight
- See also: ABCD Research Consortium. ABCD Study. Published 2015. Accessed March 20, 2022. — http://abcdstudy.org/